CLINICAL TRIAL: NCT00384891
Title: A Randomized Controlled Study Comparing Adjuvant Hyperthermia Treatment in Conjunction With Mitomycin C Versus BCG Immunotherapy (BCG) Adjuvant Treatment in Patients With Superficial Transitional Cell Carcinoma of the Bladder (STCCB)
Brief Title: Hyperthermia Treatment in Conjunction With Mitomycin C Versus Bacillus Calmette-Guérin Immunotherapy (BCG) for Superficial Bladder Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Medical Enterprises Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102.1
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Urinary Bladder Diseases; Urinary Bladder Neoplasms; Urinary Bladder Cancer; Malignant Tumor of Urinary Bladder; Urologic Diseases; Urologic Neoplasms; Neoplasms; Neoplasms by Site
Keywords: Superficial urothelial cell carcinoma of bladder; NMIBC; Non Muscle Invasive Bladder Cancer; Hyperthermia; Bladder instillation; Mitomycin C; RITE; SHTC; Intravesical
MeSH Terms: conditions — Urinary Bladder Diseases; Urinary Bladder Neoplasms; Urologic Diseases; Urologic Neoplasms; Neoplasms; Neoplasms by Site; Non-Muscle Invasive Bladder Neoplasms; Hyperthermia

ARMS (2):
- Synergo + MMC (Experimental): Combined bladder wall hyperthermia and intravesical instillation with cooled Mitomycin-C
  Interventions: Device: Synergo + MMC
- Bacillus Calmette-Guérin (Active Comparator): Intravesical instillation with BCG (Bacillus Calmette-Guérin)
  Interventions: Drug: Bacillus Calmette-Guérin

INTERVENTIONS:
Device: Synergo + MMC — Combined bladder wall hyperthermia and intravesical instillation with cooled Mitomycin-C
  Other Names: RITE; SHTC
  Arms: Synergo + MMC
Drug: Bacillus Calmette-Guérin — Intravesical instillation with BCG (Bacillus Calmette-Guérin)
  Other Names: BCG
  Arms: Bacillus Calmette-Guérin

SUMMARY:
The study is designed to compare the efficacy and safety of 2 treatment types for the prevention of tumor recurrence of superficial bladder cancer:

1. A combination of bladder wall heating and local chemotherapy (Synergo)
2. Bacillus Calmette-Guérin (BCG)

DETAILED DESCRIPTION:
The study is a randomized controlled study, designed to test the efficacy and safety of a new treatment modality for the prevention of tumor recurrence in superficial bladder cancer.

Patients must have their tumors surgically resected prior to study enrollment, and undergo a series of tests to prove their bladder is now free of tumor. Eligible patients will be randomly assigned to one of 2 treatment arms:

1. A combination of bladder wall heating and local chemotherapy (Synergo)
2. Bacillus Calmette-Guérin (BCG)

Patients will be treated during the first year of the study, and will be followed up for a total of 2 years. The follow up will include a visual evaluation of the patient's bladder by cystoscopy, a cytological examination of the urine (to look for malignant cells) and other additional exams. The patients' general welfare will be monitored through out the study.

The aim of this study is to compare the efficacy and safety of the novel treatment (Synergo) to that of the well-known BCG

ELIGIBILITY:
Inclusion Criteria:

* Superficial TCC: Any G3 or any T1 and/or CIS
* Multifocal (>1) Ta lesions
* Multiple recurrences (>2) of Ta lesions in the last 24 months
* Complete tumor eradication must be confirmed
* WHO performance status 0-2 (Appendix V)
* Life expectancy of more than 24 months
* Patients willing to sign informed consent

Exclusion Criteria:

* Bladder tumors other than TCC
* Coexistence of another primary malignant tumor other than BCC of the skin
* TCC of the bladder involving the urethra or upper urinary tract
* Previous history of TCC stage T2 or higher
* Clinical presence or previous history of regional spreading or distant metastases
* Intravesical MMC treatments during the last 12 months
* Previous intravesical BCG therapy (Any intravesical BCG therapy in the last 24 months, or More than 6 BCG intravesical instillations in the last 48 months.
* Previous pelvic radiotherapy or systemic chemotherapy
* Partial cystectomy
* Diverticle of bladder larger than 1cm in diameter
* Residual urine > 100cc measured by uroflowmetry
* Bladder volume < 150cc measured by ultrasound
* Urinary incontinence (more than one wet pad a day)
* Urethral stricture impeding 20F catheterization
* Urethral bleeding or persistent hematuria
* Active intractable or uncontrollable UTI
* Active tuberculosis or BCG infection
* Patients who experienced BCG life threatening sepsis
* Known allergy to MMC or BCG
* Known impaired immune response, positive HIV serology, patients receiving systemic steroids or immunosuppressive therapy
* Hematological disorders; leukocytes < 3500, platelets < 100,000
* Kidney or liver function disorders (more than 1.5 times upper normal limit)
* Pregnant or lactating women
* Patients who cannot be followed up properly or are unable to collaborate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2002-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | 2 years
  Recurrence free survival probability of STCCB in patients with pure (non-CIS) papillary tumor

SECONDARY OUTCOMES:
Proportion of complete response in CIS patients | 3 months
Progression rate (to disease stage>T1) and/or metastatic disease | 2 years
Local and systemic side effects, both subjective and objective | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alfred A Witjes, MD PhD, Principal Investigator — Department of Urology, Radboud University Hospital, Nijmegen, The Netherlands
Locations (8):
- University Hospital - AKH Vienna, Vienna, Austria
- Israel (3):
  - Bnai Zion Medical Center, Haifa
  - Wolfson Hospital, Holon
  - Hadassah University Hospital, Jerusalem
- Italy (3):
  - Galliera Hospital, Genova
  - Istituto Europeo del Oncologia, Milan
  - San Raffaele Hospital (HSR), Milan
- Department of Urology, Radboud University Hospital, Nijmegen, Netherlands

REFERENCES:
- [Derived] Arends TJ, Nativ O, Maffezzini M, de Cobelli O, Canepa G, Verweij F, Moskovitz B, van der Heijden AG, Witjes JA. Results of a Randomised Controlled Trial Comparing Intravesical Chemohyperthermia with Mitomycin C Versus Bacillus Calmette-Guerin for Adjuvant Treatment of Patients with Intermediate- and High-risk Non-Muscle-invasive Bladder Cancer. Eur Urol. 2016 Jun;69(6):1046-52. doi: 10.1016/j.eururo.2016.01.006. Epub 2016 Jan 20. PMID 26803476